CLINICAL TRIAL: NCT05248139
Title: Safety and Effectiveness of Single-dose Subconjunctival Triamcinolone Compared to Topical Prednisolone Eye Drops in Manual Small Incision Cataract Surgery
Brief Title: Safety and Effectiveness of Drop-free Small Incision Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Visualiza (Other)
Collaborators: Seva Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dropfree MSICS
Record Dates: First submitted 2021-12-08; First posted 2022-02-21 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Cataract; Ocular Inflammation; Ocular Hypertension; Post-Op Complication
MeSH Terms: conditions — Cataract; Ocular Hypertension; Postoperative Complications | interventions — Triamcinolone Acetonide; Triamcinolone; prednisolone acetate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-dose steroid medication delivered during surgery (Experimental): Subconjunctival injection of Triamcinolone acetonide.
  Interventions: Drug: Intraoperative delivery of medication, Kenalog (Triamcinolone)
- Standard of care post-operative steroid drops (Active Comparator): Prednisolone acetate ophthalmic solution, 4-week taper.
  Interventions: Drug: Topical post-operative eyedrops, Prednisolone acetate

INTERVENTIONS:
Drug: Intraoperative delivery of medication, Kenalog (Triamcinolone) — Subconjunctival triamcinolone acetonide 4 mg (0.4 mL of 10 mg/mL solution), single-dose injected 6-8 mm inferior to the inferior limbus with a bent 27-gauge needle at completion of cataract surgery.
  Arms: Single-dose steroid medication delivered during surgery
Drug: Topical post-operative eyedrops, Prednisolone acetate — Standard of care Presnisolone acetate 1% ophthalmic drop taper: 4 times per day for first week, then tapering one drop per week for 3 additional weeks. Discontinued after 4 weeks.
  Arms: Standard of care post-operative steroid drops

SUMMARY:
This is a randomized control trial comparing the effects of subconjunctival triamcinolone administration during surgery to topical prednisolone drops on the development of post-operative inflammation and macular edema in manual small incision cataract surgery.

DETAILED DESCRIPTION:
Eye drops given following cataract surgery for prevention of post-operative inflammation carry many disadvantages, such as cost and poor medication adherence. To eliminate these barriers, the emerging technique of single dose of subconjunctival triamcinolone delivered during surgery has been shown an effective and safe alternative. The goal of this study is to build on this evidence, utilizing subconjunctival triamcinolone in conjunction with a different surgical technique and population as what was previously studied. This is a randomized control trial comparing the effects of single-dose subconjunctival triamcinolone administration at the time of surgery to the standard 4-week taper of topical prednisolone drops following manual small incision cataract surgery in Guatemala. Patients will be evaluated at post-operative weeks 6 and 12 with the primary outcome variables of intraocular pressure and best corrected visual acuity. Data on presence and amount of corneal edema, anterior chamber inflammation, and development of macular edema will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a visually significant cataract: nuclear sclerotic, posterior subcapsular and/or cortical
* Best corrected visual acuity or 20/40 or worse

Exclusion Criteria:

* Axial length < 20 or > 26 mm
* Cataract which is traumatic, subluxated, or Morgagnian
* Presence of ocular comorbidity: including corneal or retinal abnormalities (corneal opacities, macular degeneration, macular scars, epiretinal membrane, retinal detachment, retinal vascular occlusion), glaucoma, ocular hypertension, glaucoma suspect (cup-to-disc ratio of 0.7 or more, history of steroid response, history of uveitis, pseudoexfoliation
* History of endophthalmitis or macular edema in the fellow eye
* Personal history of diabetes mellitus or uncontrolled hypertension
* Currently pregnant or lactating women
* Current use of systemic steroids for asthma, rheumatoid arthritis or other illness or history of steroid use by any route in the prior 3 months.
* Intraoperative complications including posterior capsular rupture, iris prolapse, zonular dialysis, retained nucleus, vitreous loss, iris trauma resulting in hemorrhage, Descemet dehiscence of more than 1 mm x 1 mm

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Mean post-operative intraocular pressure (IOP) in mmHg in each group | Pre-operative exam through post-operative month week 12
  Comparison of mean IOP in mmHg obtained by applanation between control and intervention groups at all time points
Corrected distance visual acuity (CDVA) | Pre-operative exam through post-operative week 12
  Comparison of visual acuity following refraction quantified on a the logarithm of the minimum angle of resolution (LogMAR) scale with a range from -0.30 (Snellen equivalent 6/3) with exceptional vision to +3.00 which corresponds to poor vision or only able to discriminate hand motions.

SECONDARY OUTCOMES:
Degree of inflammation using anterior chamber (AC) inflammation score | Pre-operative exam through post-operative week 12
  Comparison between groups; score obtained by slit lamp examination by a single, non-operating investigational surgeon at all clinic time points. Patients will receive a number for anterior chamber cell ranging from 0 which equals no inflammatory cells visible to 4, or >50 visible cells in the anterior chamber according to the Standardization of Uveitis Nomenclature (SUN) scoring system. This will then be added to the patient's flare score ranging from 0, or no flare, to 4+, which signifies high levels of inflammation, such as fixed or plastic anterior chamber fluid. The summation of these values will determine the patient's overall anterior inflammation score for that examination date.
Incidence of treatment-emergent macular edema | Post-operative month one through post-operative week 12
  Incidence of macular edema compared between treatment groups. Macular edema defined as BCVA of 20/40 or worse and ocular coherence tomography with identifiable cystoid spaces within the macula (central 1 mm) or central subfield thickening of 320 µm or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Shorstein, MD, Study Chair — Seva Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papa-Vettorazzi R, Shorstein NH, Peterson B, Yee Melgar M, Silva Linares L, O'Brien KS. Comparison of Subconjunctival Triamcinolone with Topical Prednisolone for Routine Anti-Inflammatory Prophylaxis in Manual Small Incision Cataract Surgery: A Single-Center, Randomized Controlled Trial Pilot Protocol. Clin Ophthalmol. 2025 Jul 4;19:2091-2105. doi: 10.2147/OPTH.S527039. eCollection 2025. PMID 40630265